CLINICAL TRIAL: NCT01137682
Title: A Phase III, Multicenter, Randomized, Parallel-group Study to Assess the Efficacy and Safety of Double-blind Pasireotide LAR 40 mg and Pasireotide LAR 60 mg Versus Open-label Octreotide LAR or Lanreotide ATG in Patients With Inadequately Controlled Acromegaly
Brief Title: Efficacy and Safety of Pasireotide Long Acting Release (LAR) Versus Octreotide LAR or Lanreotide Autogel (ATG) in Patients With Inadequately Controlled Acromegaly
Acronym: PAOLA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSOM230C2402; EUDRACT 2009-016722-13 (Registry Identifier: EUDRACT)
Record Dates: First submitted 2010-05-27; First posted 2010-06-04 (Estimated); Results first posted 2015-01-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Acromegaly
Keywords: Acromegaly; hormone disorder; growth hormone; insulin like growth factor-1; pituitary tumor; pasireotide; SOM230
MeSH Terms: conditions — Acromegaly; Pituitary Neoplasms | interventions — pasireotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pasireotide LAR 40 mg (Experimental): Supplied in blinded fashion as 20 and 40 mg powder in vials and 2 mL vehicle in ampoule (for reconstitution)
  Interventions: Drug: Pasireotide
- Pasireotide LAR 60 mg (Experimental): Supplied in blinded fashion as 20 and 40 mg powder in vials and 2 mL vehicle in ampoule (for reconstitution)
  Interventions: Drug: Pasireotide
- Control arm (octreotide or lanreotide) (Active Comparator): If a patient is randomized to the open label arm the investigator will either:
  * be instructed to contact a Novartis delegate to initiate shipment of either octreotide LAR 30 mg or lanreotide ATG 120 mg from a Novartis or designee depot to the site, or
  * continue to dispense either octreotide LAR 30 mg or lanreotide ATG 120 mg available at the institution to the patient if permitted by local regulations.
  Interventions: Drug: octreotide LAR 30mg; Drug: lanreotide ATG 120mg

INTERVENTIONS:
Drug: Pasireotide — * Double-blind pasireotide LAR 40 mg i.m. injection once every 28 ± 2 days for 24 weeks or
  * Double-blind pasireotide LAR 60 mg i.m. injection once every 28 ± 2 days for 24 weeks
  Other Names: SOM230
  Arms: Pasireotide LAR 40 mg; Pasireotide LAR 60 mg
Drug: octreotide LAR 30mg — In an open-label, active control arm, continue on the same treatment with octreotide LAR 30 mg every 28 ± 2 days as received for at least 6 months prior to randomization
  Arms: Control arm (octreotide or lanreotide)
Drug: lanreotide ATG 120mg — In an open-label, active control arm, continue on the same treatment with lanreotide ATG 120 mg every 28 ± 2 days as received for at least 6 months prior to randomization
  Arms: Control arm (octreotide or lanreotide)

SUMMARY:
This study will evaluate the efficacy and safety of pasireotide LAR 40 and 60 mg versus octreotide LAR or lanreotide ATG in patients with inadequately controlled acromegaly.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with written informed consent prior to any study related activity
2. Patients who had inadequately controlled acromegaly as defined by a mean GH concentration of a 5-point profile over a 2-hour period > 2.5 µg/L and sex- and age-adjusted IGF-1 > 1.3 x upper limit of normal (ULN)
3. Patients who had been treated with maximum indicated doses of octreotide LAR or lanreotide ATG for at least 6 months prior to visit 1 (screening). The maximum indicated dose for octreotide LAR was 30mg and for lanreotide ATG iwas120 mg
4. Patients who had a diagnosis of pituitary micro- or macro adenoma. Patients could have been previously submitted to surgery
5. Patients who completed the 24-week treatment period in core according to the requirements of the core study protocol or corresponding amendments could enter extension

Exclusion Criteria:

1. Patients who had received pasireotide (SOM 230) prior to enrolment
2. Concomitant treatment with Growth Hormone Receptor (GHR)-antagonist or dopamine agonists unless concomitant treatment was discontinued 8 weeks prior to visit 1 (screening)(8 weeks wash out period). Such patients must have been treated with octreotide LAR 30 mg or lanreotide ATG 120 mg monotherapy continuously for a minimum of 6 months prior to starting combination therapy and they should have been inadequately controlled on monotherapy.
3. Patients who had compression of the optic chiasm causing acute clinically significant visual field defects
4. Patients who required a surgical intervention for relief of any sign or symptom associated with tumor compression
5. Patients who had received pituitary irradiation within 10 years prior to visit 1 (screening).
6. Patients who had undergone major surgery/surgical therapy for any cause within 4 weeks prior to visit 1 (screening).
7. Patients who were hypothyroid and not adequately treated with a stable dose of thyroid hormone replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2010-07-19 (Actual); Primary Completion 2013-01-22 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (58):
- United States (4):
  - University of Michigan, Ann Arbor, Michigan
  - Oregon Health & Science University, Portland, Oregon
  - University of Texas Southwestern Medical Center Division of Hematology/Oncolog, Dallas, Texas
  - Swedish Neuroscience Institute 550 17th Avenue, Suite 500, Seattle, Washington
- Novartis Investigative Site, CABA, Buenos Aires, Argentina
- Belgium (4):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Brazil (7):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, São Luís, Maranhão
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Joinville, Santa Catarina
  - Novartis Investigative Site, Botucatu, São Paulo
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Sherbrooke, Quebec, Canada
- Colombia (3):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cali
- France (10):
  - Novartis Investigative Site, Toulouse, Cedex 9
  - Novartis Investigative Site, Bron, Cedex
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Saint Herblain - Nantes
- Germany (4):
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Petah Tikva, Israel
- Italy (5):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Napoli
- Norway (2):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo
- Poland (3):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Bucharest, Romania
- Russia (3):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Tyumen
- Saudi Arabia (2):
  - Novartis Investigative Site, Jeddah
  - Novartis Investigative Site, Riyadh
- Spain (3):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Alicante, Valencia
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Altunizade
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Izmir
- Novartis Investigative Site, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Colao A, Bronstein MD, Brue T, De Marinis L, Fleseriu M, Guitelman M, Raverot G, Shimon I, Fleck J, Gupta P, Pedroncelli AM, Gadelha MR. Pasireotide for acromegaly: long-term outcomes from an extension to the Phase III PAOLA study. Eur J Endocrinol. 2020 Jun;182(6):583. doi: 10.1530/EJE-19-0762. PMID 32217809
- [Derived] Gadelha MR, Bronstein MD, Brue T, Coculescu M, Fleseriu M, Guitelman M, Pronin V, Raverot G, Shimon I, Lievre KK, Fleck J, Aout M, Pedroncelli AM, Colao A; Pasireotide C2402 Study Group. Pasireotide versus continued treatment with octreotide or lanreotide in patients with inadequately controlled acromegaly (PAOLA): a randomised, phase 3 trial. Lancet Diabetes Endocrinol. 2014 Nov;2(11):875-84. doi: 10.1016/S2213-8587(14)70169-X. Epub 2014 Sep 24. PMID 25260838

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred ninety-eight patients were randomized and 5 patients in CORE and 1 patient in extension did not receive any study treatment
Groups:
- Pasireotide LAR 40 mg; Pasireotide LAR 60 mg: Supplied in blinded fashion as 20 and 40 mg powder in vials and 2 mL vehicle in ampoule (for reconstitution) for intramuscular administration every 28 days
- Control Arm (Octreotide or Lanreotide): Open label octreotide LAR 30 mg or lanreotide ATG 120 mg supplied either locally or from designated depot. Administered intramuscular every 28 days
Period: Overall Study
Arm/Group | Pasireotide LAR 40 mg | Pasireotide LAR 60 mg | Control Arm (Octreotide or Lanreotide)
Started | 65 | 65 | 68
Not Treated | 2 | 2 | 1
Treated | 63 | 63 | 67
Completed 24-Week Core Phase | 59 | 57 | 65
Not Continuing Into Extension | 2 | 3 | 2
Continuing Into Extension | 57 | 54 | 63
Safety Set - CORE | 63 (2 patients never received drug.) | 62 (2 patients never received drug. 1 patient had no post baseline safety assement.) | 66 (2 patients never received drug.)
Safety Set - Extension | 57 | 54 | 62 (1 patient did not receive study treatment)
Completed | 28 | 25 | 34
Not Completed | 37 | 40 | 34
Not completed — Adverse Event-CORE | 2 | 4 | 0
Not completed — Withdrawal by Subject-CORE | 2 | 2 | 2
Not completed — Administrative problems-CORE | 2 | 1 | 0
Not completed — Protocol Violation-CORE | 0 | 1 | 1
Not completed — Adverse Event-Extension | 4 | 8 | 7
Not completed — Lack of Efficacy-Extension | 15 | 9 | 13
Not completed — Withdrawal by Subject-Extension | 6 | 8 | 8
Not completed — Lost to Follow Up-Extension | 0 | 1 | 0
Not completed — Administrative problems-Extension | 0 | 2 | 0
Not completed — Death-Extension | 2 | 0 | 0
Not completed — Protocol Violation-Extension | 2 | 1 | 0
Not completed — Did not enter extension | 2 | 3 | 2
Not completed — Did not receive treatment in extension | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pasireotide LAR 40 mg | Pasireotide LAR 60 mg | Control Arm (Octreotide or Lanreotide) | Total
Number analyzed (Participants) | 65 | 65 | 68 | 198
Age, Customized [Number; unit: Participants] — CORE Period
  Participants
    <65 Years | 62 | 57 | 63 | 182
    ≥ 65 Years | 3 | 8 | 5 | 16
Sex: Female, Male [Count of Participants; unit: Participants] — CORE Period
  Participants
    Female | 38 | 35 | 38 | 111
    Male | 27 | 30 | 30 | 87
Race/Ethnicity, Customized [Number; unit: Participants] — CORE Period
  Participants
    Caucasian | 53 | 52 | 56 | 161
    Black | 3 | 8 | 4 | 15
    Other | 4 | 3 | 7 | 14
    Native American | 2 | 1 | 1 | 4
    Asian | 3 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Reduction of Mean GH Levels to < 2.5 µg/L and Normalization of Sex- and Age-adjusted IGF-1.
Description: The primary objective of this study was to compare the percentage of patients achieving biochemical control (defined as mean GH levels <2.5 µg/L and normalization of sex- and age- adjusted IGF-1) at 24 weeks with pasireotide LAR 40 mg and pasireotide LAR 60 mg separately versus continued treatment with octreotide LAR 30 mg or lanreotide autogel (ATG) 120 mg. The primary efficacy variable is the proportion of patients with a reduction of mean GH levels to < 2.5 µg/L and normalization of sex- and age-adjusted IGF-1 at 24 weeks.
Time Frame: At 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pasireotide LAR 40 mg | Pasireotide LAR 60 mg | Control Arm (Octreotide or Lanreotide)
Number analyzed (Participants) | 65 | 65 | 68
percentage of participants | 15.4 [7.63 to 26.48] | 20.0 [11.10 to 31.77] | 0 [0 to 5.28]
Statistical Analysis 1: Comparison: Pasireotide LAR 40 mg vs Control Arm (Octreotide or Lanreotide); Test type: Superiority; p = 0.0006, Regression, Logistic; An exact logistic regression model that adjusts for the randomization stratification factors was used to test the null hypothesis; Odds Ratio (OR) = 16.63, 95% CI 2-sided [lower limit 3.32] (infinity)
Statistical Analysis 2: Comparison: Pasireotide LAR 60 mg vs Control Arm (Octreotide or Lanreotide); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 23.03, 95% CI 2-sided [lower limit 4.72] (infinity)

2. Secondary Outcome: Percentage of Patients With Mean GH < 2.5 μg/L and Normalization of IGF-1, Treated With Pasireotide LAR Alone or With Concomitant Medications Used to Treat Acromegaly (Extension Full Analysis Set)
Description: The percentage of patients achieving mean growth hormone (GH) levels < 2.5 μg/L and normalization of sex and age-adjusted IGF-1 was calculated with two sided 95% confidence interval. All GH assessments were based on a 5-point mean growth hormone (GH) assessed from a 2-hour profile. Scheduled time points for blood sampling were pre-dose at 0, 30, 60, 90 and 120 minutes. Total insulin-like growth factor (IGF-1) levels were assessed with one pre-dose sample at the same visits as GH. Concomitant medication known to affect GH or IGF-1 levels were allowed in patients who were not biochemically controlled after at least one year treatment with pasireotide LAR monotherapy: dopamine agonists and growth hormone receptor antagonists (extension full analysis set)
Time Frame: Extension baseline up to approximately week 268
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pasireotide LAR 40 mg Extension: If controlled on 40 mg in CORE, remain on blinded 40 mg in extension. If patient became uncontrolled, switch to open label 60 mg
- Pasireotide LAR 60 mg Extension: If controlled on 60 mg in CORE, remain on blinded 60 mg in extension. If patient became uncontrolled, switch to open label 60 mg
- Cross Over to Pasireotide Extension: Open - label 60 mg pasireotide. Control group from CORE discontinued study if controlled in CORE. If uncontrolled in CORE, switched to open label 60 mg pasireotide. Extension blinded 40 and 60 mg switched to open label if became uncontrolled.
Arm/Group | Pasireotide LAR 40 mg Extension | Pasireotide LAR 60 mg Extension | Cross Over to Pasireotide Extension
Number analyzed (Participants) | 57 | 54 | 62
percentage of participants
  Week 16 | 19.3 [10.05 to 31.91] | 25.9 [14.96 to 39.65] | 19.4 [10.42 to 31.37]
  Week 28 | 17.5 [8.75 to 29.91] | 25.9 [14.96 to 39.65] | 19.4 [10.42 to 31.37]
  Week 40 | 21.1 [11.38 to 33.89] | 27.8 [16.46 to 41.64] | 17.7 [9.20 to 29.53]
  Week 52 | 21.1 [11.38 to 33.89] | 29.6 [17.98 to 43.61] | 21.0 [11.66 to 33.18]
  Week 64 | 22.8 [12.74 to 35.84] | 20.4 [10.63 to 33.53] | 25.8 [15.53 to 38.50]
  Week 76 | 21.1 [11.38 to 33.89] | 29.6 [17.98 to 43.61] | 27.4 [16.85 to 40.23]
  Week 88 | 24.6 [14.13 to 37.76] | 31.5 [19.52 to 45.55] | 25.8 [15.53 to 38.50]
  Week 100 | 24.6 [14.13 to 37.76] | 24.1 [13.49 to 37.64] | 32.3 [20.94 to 45.34]
  Week 112 | 24.6 [14.13 to 37.76] | 25.9 [14.96 to 39.65] | 25.8 [15.53 to 38.50]
  Week 124 | 21.1 [11.38 to 33.89] | 24.1 [13.49 to 37.64] | 25.8 [15.53 to 38.50]
  Week 136 | 15.8 [7.48 to 27.87] | 24.1 [13.49 to 37.64] | 29.0 [18.20 to 41.95]
  Week 148 | 21.1 [11.38 to 33.89] | 20.4 [10.63 to 33.53] | 29.0 [18.20 to 41.95]
  Week 160 | 19.3 [10.05 to 31.91] | 20.4 [10.63 to 33.53] | 30.6 [19.56 to 43.65]
  Week 172 | 22.8 [12.74 to 35.84] | 20.4 [10.63 to 33.53] | 21.0 [11.66 to 33.18]
  Week 184 | 17.5 [8.75 to 29.91] | 20.4 [10.63 to 33.53] | 17.7 [9.20 to 29.53]
  Week 196 | 15.8 [7.48 to 27.87] | 20.4 [10.63 to 33.53] | 24.2 [14.22 to 36.74]
  Week 208 | 17.5 [8.75 to 29.91] | 18.5 [9.25 to 31.43] | 19.4 [10.42 to 31.37]
  Week 220 | 21.1 [11.38 to 33.89] | 11.1 [4.19 to 22.63] | 14.5 [6.86 to 25.78]
  Week 232 | 14.0 [6.26 to 25.79] | 14.8 [6.62 to 27.12] | 14.5 [6.86 to 25.78]
  Week 244 | 14.0 [6.26 to 25.79] | 7.4 [2.06 to 17.89] | 11.3 [4.66 to 21.89]
  Week 256 | 10.5 [3.96 to 21.52] | 7.4 [2.06 to 17.89] | 3.2 [0.39 to 11.17]
  Week 268 | 5.3 [1.10 to 14.62] | 5.6 [1.16 to 15.39] | 1.6 [0.04 to 8.66]

3. Secondary Outcome: Percentage of Participants With Normalization of Sex- and Age-adjusted IGF-1treated With Pasireotide LAR Alone or With Concomitant Medications Used to Treat Acromegaly (Extension Full Analysis Set).
Description: The percentage of patients achieving normalization of sex and age-adjusted IGF-1 was calculated with two sided 95% confidence interval. Total insulin-like growth factor (IGF-1) levels were assessed with one pre-dose sample at the same visits as GH. Concomitant medication known to affect IGF-1 levels were allowed in patients who were not biochemically controlled after at least one year treatment with pasireotide LAR monotherapy: dopamine agonists and growth hormone receptor antagonists (Extension full analysis set)
Time Frame: Extension baseline up to approximately week 268
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pasireotide LAR 40 mg Extension | Pasireotide LAR 60 mg Extension | Cross Over to Pasireotide Extension
Number analyzed (Participants) | 57 | 54 | 62
percentage of participants
  Week 16 | 33.3 [21.40 to 47.06] | 29.0 [17.98 to 43.61] | 25.8 [15.53 to 38.50]
  Week 28 | 29.8 [18.43 to 43.40] | 33.3 [21.09 to 47.47] | 22.6 [12.93 to 34.97]
  Week 40 | 36.8 [24.45 to 50.66] | 37.0 [24.29 to 51.26] | 24.2 [14.22 to 36.74]
  Week 52 | 28.1 [16.97 to 41.54] | 33.3 [21.09 to 47.47] | 25.8 [15.53 to 38.50]
  Week 64 | 33.3 [21.40 to 47.06] | 27.8 [16.46 to 41.64] | 29.0 [18.20 to 41.95]
  Week 76 | 26.3 [15.54 to 39.66] | 35.2 [22.68 to 49.38] | 29.0 [18.20 to 41.95]
  Week 88 | 28.1 [16.97 to 41.54] | 35.2 [22.68 to 49.38] | 25.8 [15.53 to 38.50]
  Week 100 | 31.6 [19.91 to 45.24] | 29.6 [17.98 to 43.61] | 32.3 [20.94 to 45.34]
  Week 112 | 31.6 [19.91 to 45.24] | 27.8 [16.46 to 41.64] | 30.6 [19.56 to 43.65]
  Week 124 | 24.6 [14.13 to 37.76] | 31.5 [19.52 to 45.55] | 29.0 [18.20 to 41.95]
  Week 136 | 21.1 [11.38 to 33.89] | 25.9 [14.96 to 39.65] | 37.1 [25.16 to 50.31]
  Week 148 | 26.3 [15.54 to 39.66] | 22.2 [12.04 to 35.60] | 33.9 [22.33 to 47.01]
  Week 160 | 24.6 [14.13 to 37.76] | 25.9 [14.96 to 39.65] | 33.9 [22.33 to 47.01]
  Week 172 | 26.3 [15.54 to 39.66] | 22.2 [12.04 to 35.60] | 22.6 [12.93 to 34.97]
  Week 184 | 19.3 [10.05 to 31.91] | 22.2 [12.04 to 35.60] | 22.6 [12.93 to 34.97]
  Week 196 | 24.6 [14.13 to 37.76] | 22.2 [12.04 to 35.60] | 27.4 [16.85 to 40.23]
  Week 208 | 22.8 [12.74 to 35.84] | 22.2 [12.04 to 35.60] | 21.0 [11.66 to 33.18]
  Week 220 | 22.8 [12.74 to 35.84] | 11.1 [4.19 to 22.63] | 19.4 [10.42 to 31.37]
  Week 232 | 14.0 [6.26 to 25.79] | 14.8 [6.62 to 27.12] | 17.7 [9.20 to 29.53]
  Week 244 | 14.0 [6.26 to 25.79] | 9.3 [3.08 to 20.30] | 14.5 [6.86 to 25.78]
  Week 256 | 12.3 [5.08 to 23.68] | 7.4 [2.06 to 17.89] | 6.5 [1.79 to 15.70]
  Week 268 | 5.3 [1.10 to 14.62] | 5.6 [1.16 to 15.39] | 1.6 [0.04 to 8.66]

4. Secondary Outcome: Percentage of Patients With Mean GH < 2.5 μg/L Treated With Pasireotide LAR Alone or With Concomitant Medications Used to Treat Acromegaly (Extension Full Analysis Set)
Description: The percentage of patients achieving mean growth hormone (GH) levels < 2.5 μg/L was calculated with two sided 95% confidence interval. All GH assessments were based on a 5-point mean growth hormone (GH) assessed from a 2-hour profile. Scheduled time points for blood sampling were pre-dose at 0, 30, 60, 90 and 120 minutes. Concomitant medication known to affect GH levels were allowed in patients who were not biochemically controlled after at least one year treatment with pasireotide LAR monotherapy: dopamine agonists and growth hormone receptor antagonists (Extension full analysis set)
Time Frame: Extension baseline up to approximately week 268
Population: Full analysis set (FAS): comprised all patients who were randomized. Following the intent-to-treat principle, patients were analyzed according to the study drug they were assigned to at randomization and actual stratum.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Control Arm (Octreotide or Lanreotide) Extension: Open - label 60 mg pasireotide. Control group from CORE discontinued study if controlled in CORE. If uncontrolled in CORE, switched to open label 60 mg pasireotide. Extension blinded 40 and 60 mg switched to open label if became uncontrolled
Arm/Group | Pasireotide LAR 40 mg Extension | Pasireotide LAR 60 mg Extension | Control Arm (Octreotide or Lanreotide) Extension
Number analyzed (Participants) | 57 | 54 | 62
percentage of participants
  Week 16 | 38.6 [26.00 to 52.43] | 55.6 [41.40 to 69.08] | 33.9 [22.33 to 47.01]
  Week 28 | 40.4 [27.56 to 54.18] | 44.4 [30.92 to 58.60] | 43.5 [30.99 to 56.74]
  Week 40 | 38.6 [26.00 to 52.43] | 42.6 [29.23 to 56.79] | 40.3 [28.05 to 53.55]
  Week 52 | 38.6 [26.00 to 52.43] | 46.3 [32.62 to 60.39] | 41.9 [29.51 to 55.15]
  Week 64 | 40.4 [27.56 to 54.18] | 37.0 [24.29 to 51.26] | 41.9 [29.51 to 55.15]
  Week 76 | 33.3 [21.40 to 47.06] | 44.4 [30.92 to 58.60] | 45.2 [32.48 to 58.32]
  Week 88 | 40.4 [27.56 to 54.18] | 42.6 [29.23 to 56.79] | 45.2 [32.48 to 58.32]
  Week 100 | 40.4 [27.56 to 54.18] | 40.7 [27.57 to 54.97] | 46.8 [33.98 to 59.88]
  Week 112 | 36.8 [24.45 to 50.66] | 44.4 [30.92 to 58.60] | 40.3 [28.05 to 53.55]
  Week 124 | 40.4 [27.56 to 54.18] | 31.5 [19.52 to 45.55] | 41.9 [29.51 to 55.15]
  Week 136 | 36.8 [24.45 to 50.66] | 35.2 [22.68 to 49.38] | 43.5 [30.99 to 56.74]
  Week 148 | 40.4 [27.56 to 54.18] | 33.3 [21.09 to 47.47] | 43.5 [30.99 to 56.74]
  Week 160 | 38.6 [26.00 to 52.43] | 33.3 [21.09 to 47.47] | 40.3 [28.05 to 53.55]
  Week 172 | 40.4 [27.56 to 54.18] | 37.0 [24.29 to 51.26] | 38.7 [26.60 to 51.93]
  Week 184 | 33.3 [21.40 to 47.06] | 31.5 [19.52 to 45.55] | 33.9 [22.33 to 47.01]
  Week 196 | 29.8 [18.43 to 43.40] | 29.6 [17.98 to 43.61] | 35.5 [23.74 to 48.66]
  Week 208 | 31.6 [19.91 to 45.24] | 24.1 [13.49 to 37.64] | 25.8 [15.53 to 38.50]
  Week 220 | 29.8 [18.43 to 43.40] | 18.5 [9.25 to 31.43] | 22.6 [12.93 to 34.97]
  Week 232 | 24.6 [14.3 to 37.76] | 18.5 [9.25 to 31.43] | 21.0 [11.66 to 33.18]
  Week 244 | 19.3 [10.05 to 31.91] | 11.1 [4.19 to 22.63] | 12.9 [5.74 to 23.85]
  Week 256 | 15.8 [7.48 to 27.87] | 9.3 [3.08 to 20.30] | 6.5 [1.79 to 15.70]
  Week 268 | 7.0 [1.95 to 17.00] | 5.6 [1.16 to 15.39] | 3.2 [0.39 to 11.17]

5. Secondary Outcome: Percentage of Patients With Mean GH < 1.0 μg/L and Normalization of IGF-1, Treated With Pasireotide LAR Alone or With Concomitant Medications Used to Treat Acromegaly (Extension Full Analysis Set)
Description: The percentage of patients achieving mean growth hormone (GH) levels < 1.0 μg/L and normalization of sex and age-adjusted IGF-1 was calculated with two sided 95% confidence interval. All GH assessments were based on a 5-point mean growth hormone (GH) assessed from a 2-hour profile. Scheduled time points for blood sampling were pre-dose at 0, 30, 60, 90 and 120 minutes. Total insulin-like growth factor (IGF-1) levels were assessed with one pre-dose sample at the same visits as GH. Concomitant medication known to affect GH or IGF-1 levels were allowed in patients who were not biochemically controlled after at least one year treatment with pasireotide LAR monotherapy: dopamine agonists and growth hormone receptor antagonists (Extension full analysis set
Time Frame: Extension baseline up to approximately week 268
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Pasireotide LAR 40 mg Extension | Pasireotide LAR 60 mg Extension | Cross Over to Pasireotide Extension
Number analyzed (Participants) | 57 | 54 | 62
Participants
  Week 16 | 10.5 [3.96 to 21.52] | 16.7 [7.92 to 29.29] | 6.5 [1.79 to 15.70]
  Week 28 | 8.8 [2.91 to 19.30] | 14.8 [6.62 to 27.12] | 8.1 [2.67 to 17.83]
  Week 40 | 10.5 [3.96 to 21.52] | 9.3 [3.08 to 20.30] | 4.8 [1.01 to 13.50]
  Week 52 | 8.8 [2.91 to 19.30] | 13.0 [5.37 to 24.90] | 4.8 [1.01 to 13.50]
  Week 64 | 8.8 [2.91 to 19.30] | 13.0 [5.37 to 24.90] | 9.7 [3.63 to 19.88]
  Week 76 | 10.5 [3.96 to 21.52] | 13.0 [5.37 to 24.90] | 6.5 [1.79 to 15.70]
  Week 88 | 7.0 [1.95 to 17.00] | 20.4 [10.63 to 33.53] | 4.8 [1.01 to 13.50]
  Week 100 | 12.3 [5.08 to 23.68] | 14.8 [6.62 to 27.12] | 8.1 [2.67 to 17.83]
  Week 112 | 14.0 [6.26 to 25.79] | 20.4 [10.63 to 33.53] | 9.7 [3.63 to 19.88]
  Week 124 | 7.0 [1.95 to 17.00] | 14.8 [6.62 to 27.12] | 8.1 [2.67 to 17.83]
  Week 136 | 3.5 [0.43 to 12.11] | 18.5 [9.25 to 31.43] | 11.3 [4.66 to 21.89]
  Week 148 | 10.5 [3.96 to 21.52] | 14.8 [6.62 to 27.12] | 8.1 [2.67 to 17.83]
  Week 160 | 8.8 [2.91 to 19.30] | 14.8 [6.62 to 27.12] | 9.7 [3.63 to 19.88]
  Week 172 | 14.0 [6.26 to 25.79] | 13.0 [5.37 to 24.90] | 8.1 [2.67 to 17.83]
  Week 184 | 7.0 [1.95 to 17.00] | 13.0 [5.37 to 24.90] | 3.2 [0.39 to 11.17]
  Week 196 | 8.8 [2.91 to 19.30] | 13.0 [5.37 to 24.90] | 8.1 [2.67 to 17.83]
  Week 208 | 8.8 [2.91 to 19.30] | 9.3 [3.08 to 20.30] | 6.5 [1.79 to 15.70]
  Week 220 | 10.5 [3.96 to 21.52] | 7.4 [2.06 to 17.89] | 6.5 [1.79 to 15.70]
  Week 232 | 10.5 [3.96 to 21.52] | 3.7 [0.45 to 12.75] | 4.8 [1.01 to 13.50]
  Week 244 | 8.8 [2.91 to 19.30] | 3.7 [0.45 to 12.75] | 6.5 [1.79 to 15.70]
  Week 256 | 8.8 [2.91 to 19.30] | 3.7 [0.45 to 12.75] | 3.2 [0.39 to 11.17]
  Week 268 | 1.8 [0.04 to 9.39] | 3.7 [0.45 to 12.75] | 1.6 [0.04 to 8.66]

6. Secondary Outcome: Percentage of Patients With Mean GH <1.0 μg/L Treated With Pasireotide LAR Alone or With Concomitant Medications Used to Treat Acromegaly (Extension Full Analysis Set)
Description: The percentage of patients achieving mean growth hormone (GH) levels < 1.0 μg/L was calculated with two sided 95% confidence interval. All GH assessments were based on a 5-point mean growth hormone (GH) assessed from a 2-hour profile. Scheduled time points for blood sampling were pre-dose at 0, 30, 60, 90 and 120 minutes. Concomitant medication known to affect GH levels were allowed in patients who were not biochemically controlled after at least one year treatment with pasireotide LAR monotherapy: dopamine agonists and growth hormone receptor antagonists (Extension full analysis set)
Time Frame: Extension baseline up to approximately week 268
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pasireotide LAR 40 mg Extension | Pasireotide LAR 60 mg Extension | Cross Over to Pasireotide Extension
Number analyzed (Participants) | 57 | 54 | 62
percentage of participants
  Week 16 | 14.0 [6.26 to 25.79] | 27.8 [16.46 to 41.64] | 8.1 [2.67 to 17.83]
  Week 28 | 14.0 [6.26 to 25.79] | 22.2 [12.04 to 35.60] | 9.7 [3.63 to 19.88]
  Week 40 | 14.0 [6.26 to 25.79] | 13.0 [5.37 to 24.90] | 4.8 [1.01 to 13.50]
  Week 52 | 12.3 [5.08 to 23.68] | 22.2 [12.04 to 35.60] | 9.7 [3.63 to 19.88]
  Week 64 | 15.8 [7.48 to 27.87] | 18.5 [9.25 to 31.43] | 11.3 [4.66 to 21.89]
  Week 76 | 12.3 [5.08 to 23.68] | 22.2 [12.04 to 35.60] | 11.3 [4.66 to 21.89]
  Week 88 | 15.8 [7.48 to 27.87] | 22.2 [12.04 to 35.60] | 11.3 [4.66 to 21.89]
  Week 100 | 17.5 [8.75 to 29.91] | 20.4 [10.63 to 33.53] | 17.7 [9.20 to 29.53]
  Week 112 | 17.5 [8.75 to 29.91] | 25.9 [14.96 to 39.65] | 16.1 [8.02 to 27.67]
  Week 124 | 12.3 [5.08 to 23.68] | 16.7 [7.92 to 29.29] | 14.5 [6.86 to 25.78]
  Week 136 | 8.8 [2.91 to 19.30] | 25.9 [14.96 to 39.65] | 14.5 [6.86 to 25.78]
  Week 148 | 14.0 [6.26 to 25.79] | 16.7 [7.92 to 29.29] | 14.5 [6.86 to 25.78]
  Week 160 | 17.5 [8.75 to 29.91] | 18.5 [9.25 to 31.43] | 14.5 [6.86 to 25.78]
  Week 172 | 17.5 [8.75 to 29.91] | 14.8 [6.62 to 27.12] | 14.5 [6.86 to 25.78]
  Week 184 | 17.5 [8.75 to 29.91] | 18.5 [9.25 to 31.43] | 6.5 [1.79 to 15.70]
  Week 196 | 15.8 [7.48 to 27.87] | 13.0 [5.37 to 24.90] | 12.9 [5.74 to 23.85]
  Week 208 | 17.5 [8.75 to 29.91] | 13.0 [5.37 to 24.90] | 9.7 [3.63 to 19.88]
  Week 220 | 15.8 [7.48 to 27.87] | 11.1 [4.19 to 22.63] | 9.7 [3.63 to 19.88]
  Week 232 | 15.8 [7.48 to 27.87] | 3.7 [0.45 to 12.75] | 8.1 [2.67 to 17.83]
  Week 244 | 12.3 [5.08 to 23.68] | 5.6 [1.16 to 15.39] | 8.1 [2.67 to 17.83]
  Week 256 | 12.3 [5.08 to 23.68] | 3.7 [0.45 to 12.75] | 4.8 [1.01 to 13.50]
  Week 268 | 3.5 [0.43 to 12.11] | 3.7 [0.45 to 12.75] | 1.6 [0.04 to 8.66]

7. Secondary Outcome: Change From Baseline in Mean GH Values for Patients Treated With Pasireotide LAR Alone or With Concomitant Medications Used to Treat Acromegaly for CORE Visits (Extension Full Analysis Set)
Time Frame: CORE baseline up to approximately 24 weeks
Population: Number analyzed is based on available data at specific visits
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Pasireotide LAR 40 mg | Pasireotide LAR 60 mg
Number analyzed (Participants) | 57 | 54
mcg/L
  Week 12 - CORE: number analyzed (Participants) | 57 | 52
  Week 12 - CORE | -0.8 (29.77) | -6.4 (14.35)
  Week 24 - CORE: number analyzed (Participants) | 54 | 48
  Week 24 - CORE | -0.6 (32.38) | -7.2 (15.19)

8. Secondary Outcome: Change From Baseline in Mean GH Values for Patients Treated With Pasireotide LAR Alone or With Concomitant Medications Used to Treat Acromegaly for Extension Visits (Extension Full Analysis Set)
Description: Change from CORE baseline at each scheduled assessment was performed for patients randomized to pasireotide arms. Change from extension baseline at each scheduled assessment was performed for patients randomized to active control arm.
Time Frame: CORE and extension baseline up to approximately 268 weeks
Population: Available data for analysis differed from visit to visit
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Pasireotide LAR 40 mg Extension | Pasireotide LAR 60 mg Extension | Cross Over to Pasireotide Extension
Number analyzed (Participants) | 57 | 54 | 62
mcg/L
  Week 16 - extension: number analyzed (Participants) | 44 | 46 | 57
  Week 16 - extension | -7.9 (24.90) | -6.9 (14.88) | -8.4 (49.64)
  Week 28 - extension: number analyzed (Participants) | 44 | 39 | 56
  Week 28 - extension | -9.0 (24.21) | -4.5 (4.12) | -3.0 (3.86)
  Week 40 - extension: number analyzed (Participants) | 38 | 36 | 50
  Week 40 - extension | -9.7 (25.40) | -5.8 (13.93) | -11.2 (58.28)
  Week 52 - extension: number analyzed (Participants) | 36 | 35 | 46
  Week 52 - extension | -10.7 (26.60) | -7.1 (17.08) | -2.5 (3.02)
  Week 64 - extension: number analyzed (Participants) | 37 | 33 | 39
  Week 64 - extension | -11.3 (28.37) | -7.9 (17.30) | -15.7 (76.06)
  Week 76 - extension: number analyzed (Participants) | 32 | 36 | 42
  Week 76 - extension | -5.5 (5.96) | -7.2 (16.16) | -3.5 (4.27)
  Week 88 - extension: number analyzed (Participants) | 32 | 32 | 40
  Week 88 - extension | -5.7 (6.21) | -6.2 (8.55) | -3.6 (3.22)
  Week 100 - extension: number analyzed (Participants) | 34 | 31 | 39
  Week 100 - extension | -5.6 (5.71) | -5.3 (5.06) | -3.8 (4.28)
  Week 112 - extension: number analyzed (Participants) | 30 | 32 | 35
  Week 112 - extension | -5.8 (6.03) | -4.4 (6.57) | -3.9 (5.13)
  Week 124 - extension: number analyzed (Participants) | 30 | 26 | 35
  Week 124 - extension | -5.5 (5.85) | -6.0 (6.26) | -4.0 (4.36)
  Week 136 - extension: number analyzed (Participants) | 28 | 26 | 36
  Week 136 - extension | -6.0 (6.59) | -5.3 (4.99) | -4.0 (4.44)
  Week 148 - extension: number analyzed (Participants) | 29 | 25 | 35
  Week 148 - extension | -6.3 (6.21) | 6.1 (6.28) | -3.8 (3.11)
  Week 160 - extension: number analyzed (Participants) | 29 | 26 | 33
  Week 160 - extension | -5.5 (4.70) | -4.9 (5.33) | -3.2 (2.25)
  Week 172 - extension: number analyzed (Participants) | 27 | 26 | 31
  Week 172 - extension | -6.3 (6.34) | -5.9 (5.97) | -3.0 (2.47)
  Week 184 - extension: number analyzed (Participants) | 23 | 25 | 29
  Week 184 - extension | -6.3 (5.44) | -5.8 (5.79) | -3.3 (2.31)
  Week 196 - extension: number analyzed (Participants) | 22 | 21 | 29
  Week 196 - extension | -7.1 (6.81) | -6.5 (7.17) | -3.4 (2.71)
  Week 208 - extension (n=22,20,23): number analyzed (Participants) | 22 | 20 | 23
  Week 208 - extension (n=22,20,23) | -7.0 (6.82) | -6.2 (6.22) | -3.5 (2.50)
  Week 220 - extension: number analyzed (Participants) | 20 | 14 | 20
  Week 220 - extension | -7.1 (6.91) | -7.1 (8.12) | -3.8 (2.48)
  Week 232 - extension: number analyzed (Participants) | 16 | 15 | 14
  Week 232 - extension | -5.7 (5.46) | -6.8 (8.10) | -4.2 (2.46)
  Week 244 - extension: number analyzed (Participants) | 12 | 7 | 11
  Week 244 - extension | -6.0 (6.03) | -2.4 (0.90) | -4.2 (2.58)
  Week 256 - extension: number analyzed (Participants) | 10 | 6 | 6
  Week 256 - extension | -6.4 (5.91) | -4.9 (3.49) | -5.0 (3.26)
  Week 268 - extension: number analyzed (Participants) | 4 | 3 | 3
  Week 268 - extension | -3.6 (1.58) | -2.5 (0.57) | -3.7 (2.23)

9. Secondary Outcome: Change From Baseline in Standardized IGF-1 Values for Patients Treated With Pasireotide LAR Alone or With Concomitant Medications Used to Treat Acromegaly for CORE Visits (Extension Full Analysis Set)
Description: Standardized IGF-1 = IGF-1 value / ULN, where ULN is the upper limit of the normal range
Time Frame: CORE baseline up to approximately 24 weeks
Population: Available data for analysis varies from visit to visit
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Pasireotide LAR 40 mg | Pasireotide LAR 60 mg
Number analyzed (Participants) | 57 | 54
mcg/L
  CORE Week 12: number analyzed (Participants) | 57 | 53
  CORE Week 12 | 0.7 (0.97) | -1.1 (1.03)
  CORE Week 24: number analyzed (Participants) | 56 | 49
  CORE Week 24 | -0.7 (0.97) | -1.1 (1.12)

10. Secondary Outcome: Change From Baseline in Standardized IGF-1 Values for Patients Treated With Pasireotide LAR Alone or With Concomitant Medications Used to Treat Acromegaly for Extension Visits (Extension Full Analysis Set)
Description: Change from CORE baseline at each scheduled assessment was performed for patients randomized to pasireotide arms. Change from extension baseline at each scheduled assessment was performed for patients randomized to active control arm. Standardized IGF-1 = IGF-1 value / ULN, where ULN is the upper limit of the normal range
Time Frame: CORE and extension baseline up to approximately 268 weeks
Population: Available data for analysis differed from visit to visit
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Pasireotide LAR 40 mg Extension | Pasireotide LAR 60 mg Extension | Cross Over to Pasireotide Extension
Number analyzed (Participants) | 57 | 54 | 62
mcg/L
  Week 16 extension: number analyzed (Participants) | 49 | 47 | 61
  Week 16 extension | -0.8 (0.99) | -1.4 (0.97) | -0.9 (0.81)
  Week 28 extension: number analyzed (Participants) | 45 | 39 | 58
  Week 28 extension | -0.9 (1.00) | -1.3 (1.13) | -0.9 (0.88)
  Week 40 extension: number analyzed (Participants) | 42 | 37 | 51
  Week 40 extension | -1.1 (0.95) | -1.4 (0.94) | -1.1 (0.91)
  Week 52 extension: number analyzed (Participants) | 39 | 37 | 46
  Week 52 extension | -1.1 (0.90) | -1.3 (0.95) | -1.1 (0.95)
  Week 64 extension: number analyzed (Participants) | 37 | 35 | 42
  Week 64 extension | -1.3 (0.99) | -1.4 (0.98) | -1.3 (0.81)
  Week 76 extension: number analyzed (Participants) | 33 | 36 | 43
  Week 76 extension | -1.3 (0.87) | -1.5 (0.94) | -1.3 (0.84)
  Week 88 extension: number analyzed (Participants) | 33 | 32 | 41
  Week 88 extension | -1.3 (0.80) | -1.6 (1.01) | -1.3 (0.90)
  Week 100 extension: number analyzed (Participants) | 32 | 32 | 40
  Week 100 extension | -1.4 (0.93) | -1.5 (0.95) | -1.3 (0.92)
  Week 112 extension: number analyzed (Participants) | 31 | 32 | 38
  Week 112 extension | -1.5 (0.87) | -1.5 (1.00) | -1.4 (0.89)
  Week 124 extension: number analyzed (Participants) | 31 | 28 | 38
  Week 124 extension | -1.4 (0.86) | -1.5 (0.95) | -1.3 (0.97)
  Week 136 extension: number analyzed (Participants) | 29 | 27 | 38
  Week 136 extension | -1.4 (0.91) | -1.7 (0.92) | -1.4 (0.86)
  Week 148 extension: number analyzed (Participants) | 28 | 26 | 36
  Week 148 extension | -1.4 (0.86) | -1.5 (0.99) | -1.3 (0.84)
  Week 160 extension: number analyzed (Participants) | 29 | 28 | 34
  Week 160 extension | -1.4 (0.90) | -1.6 (0.87) | -1.4 (0.94)
  Week 172 extension: number analyzed (Participants) | 26 | 27 | 31
  Week 172 extension | -1.5 (0.81) | -1.6 (0.97) | -1.3 (0.98)
  Week 184 extension: number analyzed (Participants) | 23 | 25 | 31
  Week 184 extension | -1.3 (0.70) | -1.5 (1.03) | -1.4 (0.93)
  Week 196 extension: number analyzed (Participants) | 23 | 22 | 29
  Week 196 extension | -1.4 (0.81) | -1.5 (1.11) | -1.3 (1.11)
  Week 208 extension: number analyzed (Participants) | 23 | 22 | 22
  Week 208 extension | -1.4 (0.79) | -1.6 (1.00) | -1.2 (0.98)
  Week 220 extension: number analyzed (Participants) | 20 | 14 | 20
  Week 220 extension | -1.4 (0.94) | -1.6 (1.06) | -1.4 (0.91)
  Week 232 extension: number analyzed (Participants) | 15 | 15 | 15
  Week 232 extension | -1.4 (0.92) | -1.5 (1.13) | -1.7 (0.82)
  Week 244 extension: number analyzed (Participants) | 12 | 8 | 11
  Week 244 extension | -1.3 (0.75) | -1.9 (1.12) | -1.5 (0.79)
  Week 256 extension: number analyzed (Participants) | 10 | 6 | 6
  Week 256 extension | -1.3 (0.58) | -1.4 (1.39) | -1.8 (0.90)
  Week 268 extension: number analyzed (Participants) | 4 | 3 | 3
  Week 268 extension | -1.4 (0.43) | -1.7 (0.39) | -1.7 (0.81)

11. Secondary Outcome: Duration of the First Response for Patients Achieving a Reduction of Mean GH Level to < 2.5 μg/L and Normalization of IGF-1 and Treated With Pasireotide LAR Alone or With Concomitant Medications Used to Treat Acromegaly (Extension Full Analysis Set)
Description: n is the number of patients achieving response criteria. The weeks correspond to duration of first response (in weeks) for patients achieving biomedical control. Median and 95% CI are derived from Kaplan-Meier curves. Kaplan-Meier estimates [95% CI] at each time point are estimates of probability of response.
Time Frame: CORE baseline up to approximately 268 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pasireotide LAR 40 mg Extension | Pasireotide LAR 60 mg Extension | Cross Over to Pasireotide Extension
Number analyzed (Participants) | 57 | 54 | 62
weeks | 29.1 [15.6 to 48.1] | 26.9 [12.7 to 48.0] | 24.9 [12.4 to 47.4]

12. Secondary Outcome: Time to First Response (Weeks) by Treatment for Patients Achieving a Reduction of Mean GH Level to < 2.5 µg/L and Normalization of IGF-1 and Treated With Pasireotide LAR Alone or With Concomitant Medications Used to Treat Acromegaly
Description: Time to first response is defined as the time from the date of first dose to the date of first occurrence of a reduction of mean GH < 2.5 µg/L and the normalization of IGF-1. The weeks correspond to time taken to achieve first mean GH < 2.5 µg/L and the normalization of IGF-1.
Time Frame: CORE baseline up to approximately 268 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pasireotide LAR 40 mg Extension | Pasireotide LAR 60 mg Extension | Cross Over to Pasireotide Extension
Number analyzed (Participants) | 57 | 54 | 62
weeks | 112.3 [76.1 to 254.1] | 65.3 [40.4 to 94.9] | 95.1 [65.3 to 156.0]

13. Secondary Outcome: Change From Baseline in AcroQoL Total Scores for Patients Treated With Pasireotide LAR Alone or With Concomitant Medications Used to Treat Acromegaly for CORE Visits(Extension Full Analysis Set)
Description: Acromegaly Quality of Life questionnaire (AcroQoL) is a validated disease specific questionnaire. It contains 22 items divided into two scales: physical aspects (8 items) and psychological aspects (14 items) which is divided in two sub-scales: physical appearance and personal relationships of the patient (seven items each). The total score and sub-scores were calculated using the following formula: ((X -Y) / 4Y) x 100, X=sum of the scores for individual items (between 1 and 5 for each item), Y=number of individual items included in above sum (i.e. 22 for the total score, 8 for the physical sub-score, 14 for the psychological sub-score, 7 for the sub-score 'appearance' and 'personal relations'). The scoring of the questionnaire was performed as specified by the instrument developers. Total scores range from 0 to 100. Higher scores represent better quality of life. If more than 25% of items are not completed, results were considered invalid.
Time Frame: CORE baseline up to approximately 24 weeks
Population: Available data available for analysis differed from visit to visit
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pasireotide LAR 40 mg | Pasireotide LAR 60 mg
Number analyzed (Participants) | 57 | 54
scores on a scale
  Week 4 CORE: number analyzed (Participants) | 55 | 52
  Week 4 CORE | 3.5 (11.28) | 2.3 (11.08)
  Week 8 CORE: number analyzed (Participants) | 54 | 52
  Week 8 CORE | 2.4 (12.97) | 2.5 (12.11)
  Week 12 CORE: number analyzed (Participants) | 53 | 50
  Week 12 CORE | 3.0 (12.41) | 1.9 (11.50)
  Week 16 CORE: number analyzed (Participants) | 55 | 52
  Week 16 CORE | 3.3 (12.99) | 6.6 (15.33)
  Week 20 CORE: number analyzed (Participants) | 56 | 50
  Week 20 CORE | 3.5 (12.89) | 4.0 (16.02)
  Week24 CORE: number analyzed (Participants) | 55 | 53
  Week24 CORE | 3.0 (16.61) | 5.4 (17.77)

14. Secondary Outcome: Change From Baseline in AcroQoL Total Scores for Patients Treated With Pasireotide LAR Alone or With Concomitant Medications Used to Treat Acromegaly for Extension Visits (Extension Full Analysis Set)
Description: as for outcome 13
Time Frame: CORE Baseline and extension baseline up to approximately 268 weeks
Population: completed and valid questionnaires at visits
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pasireotide LAR 40 mg Extension | Pasireotide LAR 60 mg Extension | Cross Over to Pasireotide Extension
Number analyzed (Participants) | 57 | 54 | 62
scores on a scale
  Week 16 extension: number analyzed (Participants) | 50 | 46 | 61
  Week 16 extension | 4.2 (16.34) | 2.9 (19.09) | 0.8 (10.22)
  Week 28 extension: number analyzed (Participants) | 46 | 40 | 54
  Week 28 extension | 5.6 (13.21) | 4.8 (16.83) | 3.3 (10.70)
  Week 40 extension: number analyzed (Participants) | 44 | 41 | 51
  Week 40 extension | 3.2 (15.78) | 2.5 (18.21) | 3.2 (10.31)
  Week 52 extension: number analyzed (Participants) | 41 | 36 | 46
  Week 52 extension | 6.1 (14.28) | 5.7 (18.69) | 4.2 (11.01)
  Week 64 extension: number analyzed (Participants) | 37 | 35 | 43
  Week 64 extension | 5.8 (13.65) | 4.2 (18.89) | 5.4 (12.12)
  Week 76 extension: number analyzed (Participants) | 31 | 36 | 42
  Week 76 extension | 7.7 (14.93) | 2.5 (19.30) | 7.7 (15.17)
  Week 88 extension: number analyzed (Participants) | 35 | 32 | 42
  Week 88 extension | 4.6 (15.11) | 5.6 (18.08) | 6.4 (10.29)
  Week 100 extension: number analyzed (Participants) | 34 | 32 | 40
  Week 100 extension | 4.3 (14.80) | 3.9 (16.91) | 5.9 (11.13)
  Week 112 extension: number analyzed (Participants) | 32 | 31 | 39
  Week 112 extension | 4.6 (15.83) | 6.5 (18.36) | 4.1 (10.35)
  Week 124 extension: number analyzed (Participants) | 28 | 30 | 37
  Week 124 extension | 5.8 (16.46) | 2.0 (17.95) | 2.0 (10.97)
  Week 136 extension: number analyzed (Participants) | 28 | 28 | 39
  Week 136 extension | 7.5 (18.72) | 5.4 (16.73) | 6.5 (11.82)
  Week 148 extension: number analyzed (Participants) | 29 | 26 | 37
  Week 148 extension | 7.6 (18.56) | 6.8 (16.65) | 5.5 (12.95)
  Week 160 extension: number analyzed (Participants) | 30 | 26 | 31
  Week 160 extension | 7.0 (19.10) | 5.1 (15.70) | 1.5 (13.36)
  Week 172 extension: number analyzed (Participants) | 28 | 26 | 31
  Week 172 extension | 4.8 (17.97) | 5.7 (17.52) | 2.1 (12.13)
  Week 184 extension: number analyzed (Participants) | 23 | 25 | 29
  Week 184 extension | 5.8 (15.31) | 5.8 (16.83) | 1.6 (12.45)
  Week 196 extension: number analyzed (Participants) | 21 | 22 | 27
  Week 196 extension | 6.1 (16.94) | 6.0 (18.58) | 3.8 (13.11)
  Week 208 extension: number analyzed (Participants) | 22 | 23 | 21
  Week 208 extension | 1.2 (13.27) | 6.2 (17.31) | 4.5 (12.62)
  Week 220 extension: number analyzed (Participants) | 19 | 16 | 21
  Week 220 extension | 4.8 (21.99) | 5.8 (17.12) | 7.3 (16.28)
  Week 232 extension: number analyzed (Participants) | 19 | 12 | 16
  Week 232 extension | 2.1 (17.51) | -0.2 (16.73) | 7.0 (15.15)
  Week 244 extension: number analyzed (Participants) | 13 | 7 | 10
  Week 244 extension | 4.5 (20.06) | 6.3 (11.05) | 3.0 (18.65)
  Week 256 extension: number analyzed (Participants) | 10 | 6 | 7
  Week 256 extension | 6.1 (25.91) | -3.0 (7.07) | 0.3 (14.08)
  Week 268 extension: number analyzed (Participants) | 4 | 3 | 3
  Week 268 extension | 0.6 (16.74) | -4.9 (4.30) | -10.6 (7.57)

15. Secondary Outcome: Summary of Pasireotide Trough Concentrations in Acromegaly Patients Following Monthly i.m. Injections of Pasireotide LAR by Incident Dose From Start of Extension Phase up to Week 196 of the Extension Phase (PK Set)
Description: PK samples were collected for those patients treated with pasireotide LAR in the core study and who continued on pasireotide LAR in the extension phase. PK samples were collected before the injection of pasireotide LAR only at weeks 112 and 196. PK samples were also collected at weeks 48 and 132 only for all patients treated with octreotide LAR 30 mg or lanreotide ATG 120 mg in the core study who started treatment with pasireotide LAR in the extension study.
  Blood samples (2.5 mL each sample) were collected to yield 1-mL plasma for analysis of pasireotide LAR oncentration.
Time Frame: Extension baseline up to approximately 196 weeks
Population: Available data for analysis varies at visits
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Pasireotide LAR 40 mg | Pasireotide LAR 60 mg
Number analyzed (Participants) | 116 | 93
mL
  Week 48: number analyzed (Participants) | 51 | 0
  Week 48 | 5.70 (3.159) |
  Week 112: number analyzed (Participants) | 25 | 72
  Week 112 | 8.66 (4.154) | 14.06 (9.807)
  Week 132: number analyzed (Participants) | 35 | 0
  Week 132 | 9.28 (5.067) |
  Week 196: number analyzed (Participants) | 21 | 65
  Week 196 | 10.32 (5.473) | 14.96 (10.210)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 268 weeks
Description: Consistent with EudraCT disclosure specifications, Novartis has reported under the Serious adverse events fields "number of deaths resulting from adverse events" all those deaths, resulting from serious adverse events that are deemed to be causally related to treatment by the investigator. The adverse events were reported on the combined CORE and extension and there were 5 patients who never received drug and 1 with no post baseline safety assessment.
Groups:
- Pasireotide LAR 40 mg: Pasireotide LAR 40 mg
- Pasireotide LAR 60 mg: Pasireotide LAR 60 mg
- Cross-over to Pasireotide: Cross-over to pasireotide
Arm/Group | Pasireotide LAR 40 mg | Pasireotide LAR 60 mg | Cross-over to Pasireotide
All-Cause Mortality (participants affected / at risk) | 2/63 | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 18/63 | 14/62 | 20/62
Other Adverse Events (participants affected / at risk) | 59/63 | 58/62 | 61/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide LAR 40 mg (N=63) | Pasireotide LAR 60 mg (N=62) | Cross-over to Pasireotide (N=62)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Cowden's disease (Congenital, familial and genetic disorders) | 0 | 0 | 1
Inner ear disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0
Drug ineffective (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 1 | 3
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Flavivirus infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Drug administration error (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pneumocephalus (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Joint arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
Maxillofacial operation (Surgical and medical procedures) | 0 | 0 | 1
Oral surgery (Surgical and medical procedures) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide LAR 40 mg (N=63) | Pasireotide LAR 60 mg (N=62) | Cross-over to Pasireotide (N=62)
Anaemia (Blood and lymphatic system disorders) | 9 | 10 | 16
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 4
Atrioventricular block first degree (Cardiac disorders) | 6 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 10 | 10 | 6
Abdominal pain upper (Gastrointestinal disorders) | 6 | 3 | 1
Constipation (Gastrointestinal disorders) | 5 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 14 | 17 | 11
Large intestine polyp (Gastrointestinal disorders) | 2 | 1 | 4
Nausea (Gastrointestinal disorders) | 7 | 7 | 3
Vomiting (Gastrointestinal disorders) | 8 | 1 | 0
Asthenia (General disorders) | 1 | 5 | 5
Fatigue (General disorders) | 4 | 4 | 2
Pyrexia (General disorders) | 7 | 1 | 2
Biliary dilatation (Hepatobiliary disorders) | 3 | 3 | 4
Cholelithiasis (Hepatobiliary disorders) | 21 | 20 | 17
Gallbladder polyp (Hepatobiliary disorders) | 4 | 3 | 1
Hepatic steatosis (Hepatobiliary disorders) | 4 | 4 | 2
Gastroenteritis (Infections and infestations) | 2 | 6 | 0
Influenza (Infections and infestations) | 9 | 9 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 1
Urinary tract infection (Infections and infestations) | 6 | 5 | 9
Viral upper respiratory tract infection (Infections and infestations) | 7 | 9 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 4 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 6
Blood glucose increased (Investigations) | 3 | 6 | 0
Insulin-like growth factor decreased (Investigations) | 2 | 4 | 2
Lipase increased (Investigations) | 4 | 1 | 4
Weight increased (Investigations) | 1 | 0 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 20 | 25 | 16
Dyslipidaemia (Metabolism and nutrition disorders) | 4 | 1 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 6 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 25 | 24 | 15
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 4 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 7 | 7 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 9 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 7 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 4
Dizziness (Nervous system disorders) | 8 | 3 | 3
Headache (Nervous system disorders) | 18 | 6 | 8
Anxiety (Psychiatric disorders) | 5 | 3 | 2
Haematuria (Renal and urinary disorders) | 7 | 2 | 0
Renal cyst (Renal and urinary disorders) | 3 | 5 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 8 | 2
Hypertension (Vascular disorders) | 7 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.